CLINICAL TRIAL: NCT01050816
Title: An Investigator Clinical Trial to Observe Effects of CHONDRON (Autologous Chondrocytes) for 12 Months in Patients With Ankle Cartilage Defect
Brief Title: Effects of CHONDRON (Autologous Chondrocytes) With Ankle Cartilage Defect
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sewon Cellontech Co., Ltd. (Industry)
Responsible Party: Gyeong Tea , Lee, Eulji General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02CON
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Results first posted 2010-05-07 (Estimated); Last update posted 2010-05-11 (Estimated); Status verified 2010-05

CONDITIONS: Articular Cartilage Defects of Ankle Joint
Keywords: articular cartilage defects; ACI; ankle joint; chondron
MeSH Terms: interventions — Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chondron implantation (Experimental): ankle cartilage defect patients who had CHONDRON transplantation
  Interventions: Procedure: Chondron(autologous chondrocyte) Implantation

INTERVENTIONS:
Procedure: Chondron(autologous chondrocyte) Implantation — * Test drug: Chondron (more than 12 million chondrocytes in 0.4ml, i.e. 1 vial)
  * Directions and dosage:
  Suspend the cells in the vial sufficiently, and implant them in the defective part, making sure that sufficient amounts are injected.
  *30 subjects participated in this open clinical trial. Those who agreed to participate voluntarily went through screening to confirm the appropriateness for the clinical trial, and then received Gel type CHONDRON (fibrin mixed autologous chondrocytes) transplantation.
  Other Names: Chondron

SUMMARY:
An open clinical trial transplanting CHONDRON (autologous chondrocytes) to ankle cartilage defect patients who are appropriate for the trial, and evaluating the validity and safety for 12 months.

DETAILED DESCRIPTION:
This clinical trial was designed to observe effects of CHONDRON (autologous chondrocytes) for 12 months in patients with ankle cartilage defects. In this clinical trial, 30 subjects were screened- 4 were excluded half way and 26 finished the trial. Full-thickness articular cartilage specimen was obtained from sites that do not have direct articulation within the ankle joint(anterior talus, anterior process of calcaneus, calcaneocuboid joint area.) Gel-type CHONDRON (Fibrin mixed Autologous chondrocytes) was transplanted at the defects. Evaluation variables were AOFAS, 100 mm VAS, HANNOVER score, self-assessment of improvement by the patient, MRI and arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

1. adult men and women over 15 and less than 65 years of age
2. applied to patients with arthroscopically or grossly confirmed, partial cartilage defect at the ankle joint
3. patients with ankle-tibia malalignment of the ankle joint, unstable ankle ligaments, bone defects at the cartilage defect area or patients who received correction in advance.
4. patients which surrounding cartilage are normal
5. patients who agreed to clinical trial participation voluntarily or by the will of the person in parental authority, and signed the written consent form

Exclusion Criteria:

1. patients hypersensitive to bovine protein
2. patients hypersensitive to gentamicin antibiotics
3. patients with inflammatory arthritis such as rheumatoid arthritis, gout arthritis
4. patients with arthritis related to autoimmune disease
5. pregnant, breast-feeding patients or those who have a possibility of pregnancy
6. patients with accompanying diseases other than articular cartilage defects, including tumors
7. patients who have a history of receiving radiotherapy, chemotherapy in the last 2 years
8. patients with diabetes (however, patients whose blood sugar test results are normal and do not have any complication of diabetes, when a written opinion that CHONDRON administration is possible is appended by a doctor are excluded)
9. patients who are administering antibiotics and antimicrobial agents due to infection
10. patients who receive steroid hormone therapy
11. Patients with psychiatric disorder and those who are considered to be inappropriate for this trial by the judgment of the clinical trial manager

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gyeung Tea Lee, MD, Principal Investigator — Eulji General Hospital
Locations (1):
- Sewon Cellontech, Seoul, Sungdong-ku, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 subjects who have ankle cartilage defects
Groups:
- Chondron Implantation: Those who agreed to participate voluntarily went through screening to confirm the appropriateness for the clinical trial, and then received appropriate amounts(by size, but mean:4vail(1.6ml)) of CHONDRON (autologous chondrocytes) transplantation.
Period: Overall Study
Arm/Group | Chondron Implantation
Started | 30
Completed | 26
Not Completed | 4
Not completed — Lost to Follow-up | 2
Not completed — patient's refusal | 2

BASELINE CHARACTERISTICS:
Arm/Group | Chondron Implantation
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 36.67 (11.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 26
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 30

OUTCOME MEASURES:

1. Primary Outcome: Average Change From Baseline in American Orthopedic Foot and Ankle Society(AOFAS) at 12 Months Post-surgery
Description: AOFAS scores(best score-100,worst score- 0 )
  1. pain-none:40/Strong and Always present:O
  2. Function
     * activities-without support activities:10/need restrain, clutch , walker or wheelchair:0
     * Maximum gait distance- more than 6:5/ less than 1:0
     * gait surface-easy in any surace:5/strong difficult in irregular ground stair or slopes:0
     * Gait abnormality-none:8/marked:0
     * saggital mobidity- normal or minimal restrain:6/strong restraint:0
     * hindfoot mobidity -normal minimal restrain:6/strong restrain:0
     * ankle and hindfoot stability - stable:8/unstable:0
  3. alignment- good:10/bad:0
Time Frame: baseline(preoperative stage),12months post-surgery
Population: Among the 30 patients, 27 who received CHONDRON transplantation became subjects for Full Analysis Set(FAS) analysis, as validity evaluation analysis subjects. The remaining 3 patients were omitted, being excluded from the FAS analysis. (1 subject refused to participate, 2 were unable to do follow-up.)
Measure: Mean (Standard Deviation); unit: scores
Arm/Group | Chondron Implantation
Number analyzed (Participants) | 27
scores | 16.93 (13.04)

2. Secondary Outcome: Average Change From Baseline in 100mm Visual Analogue Scale(VAS) at 12months Post-surgery
Description: A VAS is a horizontal line, 100mm in length, anchored by word descriptors about pain at each end.The VAS is measured degree of pain from 0mm to 100mm. Severe pain is represented by 100mm and no pain is represented by 0mm. The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks.
  The difference of secondary evaluation variables VAS at baseline and after the end of the trial were analyzed by using paired t-test. Improvements were compared and analysis by each time point.
Time Frame: baseline(preoperative stage),12months post-surgery
Population: Among the 30 patients, 27 who received CHONDRON transplantation became subjects for FAS analysis, as validity evaluation analysis subjects. The remaining 3 patients were omitted, being excluded from the FAS analysis. (1 subject refused to participate, 2 were unable to do follow-up.)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Chondron Implantation
Number analyzed (Participants) | 27
mm | -27.19 (31.33)

3. Secondary Outcome: Average Change From Baseline in the Modified Hannover Scoring System at 12 Months Post Surgery
Description: The Modified Hannover Score System contains information about patient's status(pain-36, clinical finding- 4, patient's subjective assessment- 25, statics- 6, fuction- 26, radiology-7;best score-104, worst score-0).The scores of 27 patients in the FAS group were taken in the screening period (Visit S), 12 months after transplantation (Visit 7). The difference of the scores at screening and 12 months after transplantation was compared by using the paired t-test. Improvements were compared and analyzed at each time point.
Time Frame: baseline(preoperative stage),12months post-surgery
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores
Arm/Group | Chondron Implantation
Number analyzed (Participants) | 27
scores | 26.26 (18.07)

ADVERSE EVENTS:
Time Frame: Observations are done during the screening period, on the day of cartilage sampling, CHONDRON transplantation, and 1 week, 6 week, 3 months, 6 months, and 12 months after surgery.
Description: Vital signs (blood pressure, pulse rate, body temperature) were measured on the day of sampling, transplantation, and 1 week after surgery and were recorded in the case record. Clinicopathologic tests were done in the screening period (Screening), on the days of tissue sampling and of transplantation. Results were written in the case record.
Arm/Group | Chondron Implantation
Serious Adverse Events (participants affected / at risk) | 2/30
Other Adverse Events (participants affected / at risk) | 25/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chondron Implantation (N=30)
malleolar ostoeotomy nonunion (Musculoskeletal and connective tissue disorders) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chondron Implantation (N=30)
nausea (Gastrointestinal disorders) | 8 (8)
dyspepsia (Gastrointestinal disorders) | 2 (4)
vomiting (Gastrointestinal disorders) | 2 (2)
epigastric soreness' (Gastrointestinal disorders) | 3 (3)
abdominal pain (Gastrointestinal disorders) | 2 (2)
gastritis (Gastrointestinal disorders) | 1 (1)
polyp (Gastrointestinal disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1)
defecation disorder' (Gastrointestinal disorders) | 1 (1)
pain (Musculoskeletal and connective tissue disorders) | 10 (19)
malleolar osteotomy site pain (Musculoskeletal and connective tissue disorders) | 1 (1)
lower extremities numbness (Musculoskeletal and connective tissue disorders) | 2 (2)
sholuder pain (Musculoskeletal and connective tissue disorders) | 1 (1)
lower extremities pain (Musculoskeletal and connective tissue disorders) | 1 (1)
dysuria (Renal and urinary disorders) | 2 (2)
testicular pain (Renal and urinary disorders) | 1 (1)
proteinuria (Renal and urinary disorders) | 1 (1)
edema (General disorders) | 2 (5)
headache (General disorders) | 4 (6)
Fever (General disorders) | 2 (2)
insomnia (Psychiatric disorders) | 1 (1)
vertigo (Nervous system disorders) | 1 (1)
eczema (Skin and subcutaneous tissue disorders) | 2 (2)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less